CLINICAL TRIAL: NCT04286542
Title: Identification of Mediators Associated With Presence of Nasal Hyperreactivity in Allergic Rhinitis and Chronic Rhinosinusitis
Brief Title: Mediators in Nasal Hyperreactivity in Allergic Rhinitis and Chronic Rhinosinusitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Laura Van Gerven, Professor doctor, Universitaire Ziekenhuizen KU Leuven
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: S63139
Record Dates: First submitted 2020-02-21; First posted 2020-02-27 (Actual); Last update posted 2022-05-25 (Actual); Status verified 2022-05

CONDITIONS: Hyperactivity; Allergic Rhinitis Due to House Dust Mite; Chronic Rhinosinusitis With Nasal Polyps
MeSH Terms: conditions — Spasm | interventions — Cold Temperature

STUDY DESIGN:
Intervention Model Description: Visit 1: screening, baseline sample collection. Visit 2: sample collection, provocation with cold dry air, sample collection
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Provocation with cold air (Experimental): Participants will be exposed to cold dry air for 15 minutes
  Interventions: Diagnostic Test: Cold, dry air

INTERVENTIONS:
Diagnostic Test: Cold, dry air — Participants will be exposed to cold (<-10°C, <10% relative humidity), dry air for 15 minutes.

SUMMARY:
Rhinitis, or inflammation of the nasal mucosa, can present with nasal obstruction, nasal discharge, itch or sneezing. If the sinusal mucosa is involved as well, it is called rhinosinusitis and facial pain or loss of smell is possible. Several causes are known, such as an underlying allergy ("allergic rhinitis", AR). If at least 2 symptoms are present for at least 12 weeks, it is called "chronic rhinosinusitis" (CRS).

Up to 2/3 of the AR and CRS patients have symptoms upon exposure to triggers such as sudden temperature changes, smoke, fragrances… a phenomenon called "nasal hyperreactivity" (NHR). It is currently not clear why some patients suffer NHR while others do not.

In this study, the investigators want to identify the mediators associated with NHR in patients with allergic rhinitis, chronic rhinosinusitis and healthy control subjects.To do so, participants will be provoked with cold, dry air in order to objectively diagnose NHR. Before and after provocation, the peak nasal inspiratory flow will be measured and samples will be collected (nasal secretions, biopsies).

DETAILED DESCRIPTION:
Patients with perennial allergic rhinitis, chronic rhinosinusitis with nasal polyps and healthy control subjects will be recruited. At baseline, nasal secretions and mucosal biopsies will be collected. After 3 weeks, participants will be provoked with cold, dry air, and samples will be harvested again. A decrease in the peak nasal inspiratory flow of >20% will be used as a cutoff to define nasal hyperreactivity.

Nasal secretions will be analysed for various mediators using a multiplex assay. The biopsies will be used for RT-q-PCR and immunohistochemistry of various transient receptor potential (TRP) channels.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years
* positive skin prick test for house dust mite (for allergic rhinitis group), presence of nasal polyps (for chronic rhinosinusitis with nasal polyps group)
* VAS-score >5 for rhino(sinus)itis symptoms

Exclusion Criteria:

* positive skin prick test (for chronic rhinosinusitis with nasal polyps group and healthy control group), presence of nasal polyps (for allergic rhinitis group and healthy control group)
* Acute rhinitis in the past 2 weeks
* (History of) immunotherapy for house dust mite
* Relevant anatomic abnormalities
* Participation in another clinical trial at the moment of this study.
* Use of anticoagulants (apart from acetylsalicylic acid)
* Use of tricyclic antidepressants
* History of intranasal drug usage in the past 12 months
* Pregnancy or breastfeeding
* Malignancy or severe comorbidity

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2020-01-20 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Objective nasal hyperreactivity | 3 weeks
  The peak nasal inspiratory flow will be measured before and after provocation with cold, dry air. A decrease of >20% will be used as a cutoff to objectively diagnose nasal hyperreactivity.

SECONDARY OUTCOMES:
Levels of histamine in nasal secretions | 3 weeks
  In nasal secretions, the investigators will measure the levels of histamine by using a multiplex assay. They will do so at baseline and after cold dry air provocation test.
Levels of tryptase in nasal secretions | 3 weeks
  In nasal secretions, the investigators will measure the levels of tryptase by using a multiplex assay. They will do so at baseline and after cold dry air provocation test.
Levels of substance P in nasal secretions | 3 weeks
  In nasal secretions, the investigators will measure the levels of substance P by using a multiplex assay. They will do so at baseline and after cold dry air provocation test.
Levels of neurokinin A in nasal secretions | 3 weeks
  In nasal secretions, the investigators will measure the levels of neurokinin A by using a multiplex assay. They will do so at baseline and after cold dry air provocation test.
Levels of neurokinin B in nasal secretions | 3 weeks
  In nasal secretions, the investigators will measure the levels of neurokinin B by using a multiplex assay. They will do so at baseline and after cold dry air provocation test.
Levels of calcitonin gene-related peptide in nasal secretions | 3 weeks
  In nasal secretions, the investigators will measure the levels of calcitonin gene-related peptide by using a multiplex assay. They will do so at baseline and after cold dry air provocation test.
Levels of interleukin (IL) 4 in nasal secretions | 3 weeks
  In nasal secretions, the investigators will measure the levels of IL-4 by using a multiplex assay. They will do so at baseline and after cold dry air provocation test.
Levels of IL-5 in nasal secretions | 3 weeks
  In nasal secretions, the investigators will measure the levels of IL-5 by using a multiplex assay. They will do so at baseline and after cold dry air provocation test.
Levels of IL-13 in nasal secretions | 3 weeks
  In nasal secretions, the investigators will measure the levels of IL-13 by using a multiplex assay. They will do so at baseline and after cold dry air provocation test.
Presence of TRP Vanilloid 1 in nasal mucosa. | 3 weeks
  The investigators will determine the presence of TRP vanilloid 1 on nasal mucosal biopsies at baseline and after provocation with cold, dry air by using RT-q-PCR and immunohistochemistry.
Presence of TRP Ankyrin 1 in nasal mucosa. | 3 weeks
  The investigators will determine the presence of TRP Ankyrin 1 on nasal mucosal biopsies at baseline and after provocation with cold, dry air by using RT-q-PCR and immunohistochemistry.
Presence of TRP Melastatin 8 in nasal mucosa. | 3 weeks
  The investigators will determine the presence of TRP Melastatin 8 on nasal mucosal biopsies at baseline and after provocation with cold, dry air by using RT-q-PCR and immunohistochemistry.

CONTACTS AND LOCATIONS:
Locations (1):
- KULeuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No